CLINICAL TRIAL: NCT06822023
Title: Virtual Reality and Its Use in Reducing Perioperative Stress in Cataract Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23/WS/0110
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Virtual Reality; Eye Disease; Cataract Surgery Anesthesia; Cataract Surgery
Keywords: cataract surgery, sedation, anxiety, virtual reality
MeSH Terms: conditions — Eye Diseases; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional group (No Intervention): patients will be prepared as per the standard routine; clinical and further explanation of the procedure will be given. Before proceeding to the anaesthetic room, the patients will complete the anxiety score questionnaire again and given the option to proceed with sedation or opt out.
- Interventional Group (Experimental): patients will be prepared as per the standard routine clinical care; they will then be wearing the VR mask for 10 minutes. Before proceeding to the anaesthetic room, patients will complete the anxiety score questionnaire again and given the option to proceed with sedation or opt out
  Interventions: Device: virtual reality mask

INTERVENTIONS:
Device: virtual reality mask — Patients will be prepared as per the standard routine clinical care; they will then be wearing the VR mask for 10 minutes. No other study have looked into VR mask prior to cataract surgery
  Arms: Interventional Group

SUMMARY:
This project is to evaluate the benefits of utilising virtual reality (VR) headsets with the aim of reducing peri-operative anxiety in cataract surgery and hence reducing the need for sedation in patients with significant stress levels noted during preassessment. This is a novel study, and with the increased use of VR technology throughout medicine, we may be able to offer our patients alternative management modalities to reduce stress and reduce need for medications with their subsequent potential side effects. It may also improve the quality of care provided and patients' experience with the cataract extraction procedure and might reduce the social care burden associated with standard sedation procedures. All patients will need to fill a quick preoperative anxiety and information scale questionnaire to assess their level of anxiety utilising The Amsterdam Preoperative Anxiety and Information Score.

Patients will be randomised into 2 groups:

1. Conventional group: patients will be prepared as per the standard routine clinical and further explanation of the procedure will be given. Before proceeding to the anaesthetic room, the patients will complete the anxiety score questionnaire again and given the option to proceed with sedation or opt out.
2. Interventional Group: patients will be prepared as per the standard routine clinical care; they will then be wearing the VR mask for 10 minutes. Before proceeding to the anaesthetic room, patients will complete the anxiety score questionnaire again and given the option to proceed with sedation or opt out.

Post operation, a record will be taken of the surgeon's decision on whether they want the second eye cataract surgery to be done under sedation (this is already standard practice at our centre). Finally, the patient will be asked to fill in one final grading score on whether they are happy with their decision to take/not take sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients listed for cataract surgery under local anaesthetic (topical or regional) with sedation planned.
2. First eye cataract procedures will only be included.
3. Capacity to give informed consent, cognitive and linguistic ability sufficient to understand and fill out questionnaire

Exclusion Criteria:

1. Epilepsy
2. severe vertigo
3. poor visual acuity (below 6/60 best corrected in the best seeing eye)
4. significant hearing impairment
5. recent facial injury/burn.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-12 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety score | 10 mins following intervention
  Percentage of reduction in Anxiety score in interventional group as compared to control group as assessed using the Amsterdam preoperative anxiety and information score

SECONDARY OUTCOMES:
Patient required sedation after intervention | 10 mins
  Percentage of patients who were happy with their decision to undergo/not undergo sedation in intervention vs control group.
Patient required sedation for second eye surgery | Following surgery, approximately 30-60 mins following intervention
  Percentage of patients who the surgeons would list their second eye for sedation in intervention vs control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Y Ng, MBChB, FRCOphth, Principal Investigator — south tyneside sunderland foundation trust

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jacobi PC, Dietlein TS, Jacobi FK. A comparative study of topical vs retrobulbar anesthesia in complicated cataract surgery. Arch Ophthalmol. 2000 Aug;118(8):1037-43. doi: 10.1001/archopht.118.8.1037. PMID 10922195
- See also: Cataract Statistics & Resources [Internet] — https://www.lasereyesurgeryhub.co.uk/data/cataract-statistics/